CLINICAL TRIAL: NCT00881465
Title: Videophone Administered Cognitive-Behavioral Therapy for Pediatric Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Eric Storch, Ph.D., University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USF-09-0155
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-behavioral therapy (Experimental): Cognitive-Behavioral Therapy. The psychotherapy protocol will include 14 90-minute sessions of videophone administered CBT over 12 weeks. The first session will be held face-to-face to foster rapport. Sessions 1-4 will be held twice weekly; thereafter sessions will be held weekly. Sessions 1-3 are devoted to psychoeducation, treatment discussion, and hierarchy development. Sessions 4-10 involve CBT exercises specific to each youth.
  Interventions: Behavioral: Cognitive-behavioral therapy
- Waitlist (Placebo Comparator): Waitlist Control. The participant and his/her parents will be instructed to not obtain treatment outside of the protocol or make medication changes/additions. This will be assessed through interview at the Post-Waitlist assessment.
  Interventions: Behavioral: Wait-list control

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Cognitive-Behavioral Therapy. The psychotherapy protocol will include 14 90-minute sessions of videophone administered CBT over 12 weeks.
  Arms: Cognitive-behavioral therapy
Behavioral: Wait-list control — Waitlist Control. The participant and his/her parents will be instructed to not obtain treatment outside of the protocol or make medication changes/additions. This will be assessed through interview at the Post-Waitlist assessment.
  Arms: Waitlist

SUMMARY:
Although cognitive-behavioral therapy (CBT) is the most effective intervention for pediatric obsessive-compulsive disorder (OCD), many people do receive CBT initially. Given this, alternative ways of providing CBT need to be identified and tested. With this in mind, the proposed study examines the efficacy of a videophone based cognitive-behavioral intervention for youth with OCD. A total of 30 youth will be randomly assigned to either videophone administered CBT or an abbreviated wait-list control arm. Comprehensive assessments will be conducted by trained clinicians at relevant time-points to assess symptom severity and impairment.

DETAILED DESCRIPTION:
Although cognitive-behavioral therapy (CBT) is the most effective intervention for pediatric obsessive-compulsive disorder (OCD), many people do receive CBT initially due, in part, to the lack of trained providers and geographic barriers (e.g., distance to such providers). Rather, the majority of youth with OCD receive psychiatric medication alone or together with unproven forms of psychotherapy. While some serotonergic medications have demonstrated utility in pediatric OCD, side effects can be common, response rates are modest at best, and symptom remission is rare. Given this, alternative ways of providing CBT need to be identified and tested to increase the number of people with access to this form of treatment. With this in mind, the proposed study examines the efficacy of a videophone based cognitive-behavioral intervention for youth with OCD. A total of 30 youth will be randomly assigned to either videophone administered CBT or an abbreviated wait-list control arm. Cognitive-behavioral therapy will be based on a demonstrated effective treatment protocol, and adapted for videophone administration. Comprehensive assessments will be conducted by trained clinicians at relevant time-points (e.g., baseline, post-treatment, follow-up) to assess symptom severity and impairment. Should supporting data be found, videophone-administered CBT would have the potential to help many more families who would otherwise remain untreated or inadequately treated. On a societal level, evaluation and dissemination of telehealth interventions such as this will lessen costs related to sustained treatment and OCD related impairment.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of OCD on the ADIS-IV-C/P and CY-BOCS Total Score ≥ 16
* No change in psychotropic medication (if applicable) for at least 8 weeks prior to study entry
* 7 to 17 years old
* Availability of at least one parent to accompany the child to all assessment sessions and be present for videophone sessions
* Have a computer within their home

Exclusion Criteria:

* History of and/or current psychosis, autism, bipolar disorder, or current suicidality
* Principal diagnosis other than OCD
* A positive diagnosis in the caregiver of mental retardation, psychosis, or other psychiatric disorders or conditions that would limit their ability to understand CBT (based on clinical interview)
* The child requires a higher level of psychiatric and/or medical care (e.g., inpatient hospitalization)
* Child receptive vocabulary < 80.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storch, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, St. Petersburg, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive-behavioral Therapy | Waitlist
Started | 16 | 15
Completed | 14 | 15
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-behavioral Therapy | Waitlist | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 15 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (2.5) | 11.2 (2.81) | 11.1 (2.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS; Scahill et al., 1997). The CY-BOCS is a 10-item Semi-structured Measure of Obsession and Compulsion Severity Over the Previous Week. This Measure Will Serve as the Primary Outcome Index.
Description: Items on this scale are summed to arrive at a total score. Scores on this scale range from 0 to 40 with higher scores corresponding to worse symptom severity.
Time Frame: within one week after treatment condition was concluded
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Waitlist
Number analyzed (Participants) | 16 | 15
units on a scale | 11.13 (10.53) | 18.53 (8.11)

2. Secondary Outcome: Clinical Global Impression - Severity (CGI-S; National Institute of Mental Health, 1985). The CGI-S is a 7-point Clinician Rating of Severity of Psychopathology.
Description: Scores on this scale range from 0 to 6 with higher scores corresponding to worse symptom severity.
Time Frame: within one week after treatment condition was concluded
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Waitlist
Number analyzed (Participants) | 16 | 15
units on a scale | 1.56 (1.75) | 2.47 (1.30)

3. Secondary Outcome: Clinical Global Improvement (CGI; Guy, 1976). The CGI is a 7-point Rating of Treatment Response Anchored by 1 ("Very Much Improved) and 7 ("Very Much Worse").
Description: Scores on this scale range from 1 to 7. Scores of 1 (very much improved) and 2 (much improved) are grouped together to indicate if a participate has had a beneficial response to the interview. The data represents participants who had a beneficial response to the treatment condition. Scores of 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse) and 7 (very much worse) are grouped together to indicate that a participant has not had a positive treatment response.
Time Frame: within one week after treatment condition was concluded
Measure: Number; unit: participants
Arm/Group | Cognitive-behavioral Therapy | Waitlist
Number analyzed (Participants) | 16 | 15
participants | 13 | 2

ADVERSE EVENTS:
Arm/Group | Cognitive-behavioral Therapy | Waitlist
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

LIMITATIONS AND CAVEATS:
Use of a non-active control condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes